CLINICAL TRIAL: NCT00920933
Title: Double Blind, Placebo Controlled, Parallel Group Study With an Open Label Reference Arm to Assess the Effects of Intravenously Administered AIN457 on Ozone Induced Neutrophilia Compared to Placebo & Oral Corticosteroid in Healthy Volunteers
Brief Title: Effect of AIN457 on Ozone-induced Airway Neutrophilia Compared to Placebo and Corticosteroid in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CAIN457A2104; 2008-002854-39
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Ozone challenge; airway neutrophilia; induced sputum; Healthy volunteers
MeSH Terms: interventions — secukinumab; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- AIN457 (Experimental)
  Interventions: Biological: AIN457
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- oral corticosteroid (Active Comparator)
  Interventions: Drug: prednisolone

INTERVENTIONS:
Biological: AIN457
  Arms: AIN457
Other: Placebo
  Arms: Placebo
Drug: prednisolone
  Arms: oral corticosteroid

SUMMARY:
This study will assess the ability of AIN457 to attenuate the increase in airway neutrophils that is seen following ozone exposure. Healthy subjects will be treated with AIN457, placebo, or oral corticosteroid and the response to a subsequent ozone exposure will be evaluated.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects
* Normal sputum neutrophil levels at screening
* Ozone responsive

Exclusion criteria:

* Smokers
* Prior treatment with antibody treatment or immunosuppressive agent
* Presence or history of a major chronic inflammatory autoimmune disease
* History of severe hypersensitivity to any biological agents (antibody or soluble receptor), a history of serious allergic reaction, collagen disease, neurological disease (including demyelinating disease).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Total neutrophil cell count in 106/mL in induced sputum | Day 16

SECONDARY OUTCOMES:
Serum total IL-17A | Day 1- Day 120
Percentage neutrophil cell count in induced sputum | Day 16
Safety and tolerability. Safety assessments will include vital signs, electrocardiograms (ECG), spirometry, pulse oximetry, immunogenicity and adverse events (AEs) | Day 1-Day 120
Airway function (FEV1, FVC, and FEF25-75) | 4h, 24h, and 48h after the start of the ozone exposure
Serum AIN457 pharmacokinetics (PK) | Day1-Day 120

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Großhansdorf, Germany